CLINICAL TRIAL: NCT01402622
Title: The Effect of Total Intravenous Anesthesia With Propofol on Postoperative Nausea and Vomiting in Patients Undergoing Robot-assisted Laparoscopic Radical Prostatectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sun-Joon Bai / Associate Professor, Department of Anesthesiology and Pain Medicine and Anesthesia and Pain Research Institute, Yonsei University Health System
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 4-2010-0361
Record Dates: First submitted 2011-07-25; First posted 2011-07-26 (Estimated); Last update posted 2011-07-26 (Estimated); Status verified 2011-07

CONDITIONS: Robotic Radical Prostatectomy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control group (Active Comparator): balanced anaesthesia with antiemetic prophylaxis
  Interventions: Drug: Propofol anesthesia
- TIVA group (Active Comparator): TIVA without antiemetic prophylaxis
  Interventions: Drug: Propofol anesthesia
- TIVA-P group (Active Comparator): TIVA with antiemetic prophylaxis
  Interventions: Drug: Propofol anesthesia

INTERVENTIONS:
Drug: Propofol anesthesia — In the TIVA and TIVA-P group, propofol and remifentanil were used for induction and maintenance of anaesthesia. In the control group, propofol and remifentanil were used for induction and anaesthesia was maintained with desflurane and remifentanil. In the control and TIVA-P group, ramosetron 0.3mg was administered at the end of surgery. In all patients, postoperative pain was controlled with fentanyl-based intravenous patient-controlled analgesia. he depth of anaesthesia was monitored with a bispectral index score monitor and maintained at 40-60.

SUMMARY:
To maximize the surgical visual field, Robot-assisted laparoscopic radical prostatectomy (RLRP) usually requires the patient to be positioned in a steep trendelenburg position in combination with prolonged intraperitoneal carbon dioxide (CO2) insufflation and increased intrabdominal pressure. Insufflations of CO2 during laparoscopic surgery, which causes stretch and irritation of the peritoneum, is known to play an important role in postoperative nausea and vomiting (PONV). In addition, prolonged pneumoperitoneum increases the risk for PONV. PONV can cause patient discomfort and prolong post anaesthesia care unit (PACU) stay. In addition, the patient with PONV is also predisposed to severe complications such as aspiration pneumonia, increased wound dehiscence, delayed recovery, prolonged hospital stay, and eventually increased medical cost.

DETAILED DESCRIPTION:
To maximize the surgical visual field, Robot-assisted laparoscopic radical prostatectomy (RLRP) usually requires the patient to be positioned in a steep trendelenburg position in combination with prolonged intraperitoneal carbon dioxide (CO2) insufflation and increased intrabdominal pressure. Insufflations of CO2 during laparoscopic surgery, which causes stretch and irritation of the peritoneum, is known to play an important role in postoperative nausea and vomiting (PONV). In addition, prolonged pneumoperitoneum increases the risk for PONV. PONV can cause patient discomfort and prolong post anaesthesia care unit (PACU) stay. In addition, the patient with PONV is also predisposed to severe complications such as aspiration pneumonia, increased wound dehiscence, delayed recovery, prolonged hospital stay, and eventually increased medical cost. Therefore, as RLRP itself can be an important risk factor of PONV, the anaesthesiologist should give attention to prevent PONV in this patient group, although they usually have lower risk in terms of patient-related factors. Previously published studies have recommended antiemetic prophylaxis for the patients with moderate-to-high risk of PONV. However, despite routine use of prophylactic antiemetics, laparoscopic surgery has been associated with higher incidence of PONV.Previous clinical studies suggested that total intravenous anaesthesia (TIVA) with propofol reduced PONV significantly compared to inhaled anaesthetics. Also, several studies have recommended TIVA with propofol as the anaesthetic method in patients with high risk of PONV. However none of these studies were designed and powered to detect differences in PONV in patients undergoing laparoscopic surgery, especially RLRP.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing RLRP, ASA physical status I or II, age 50 to 70.

Exclusion Criteria:

* Emergency operation.
* patients with motion sickness or PONV history to control anticipated risk of PONV.
* Patients with antiemetic use within 24 hours before surgery.
* Patients with regular corticosteroid use.
* Patients with chemotherapy within 4 or radiotherapy within 8 weeks.
* Patients with allergy to any of the study drugs.
* Patients with liver dysfunction, confirmed renal impairment, or obesity (body mass index > 35 kg/m2).

Ages: 50 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2010-12; Primary Completion 2011-04 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
the incidence and severity of PONV(Postoperative nausea and vomiting) | 48 hours after the surgery
  Comparison of the incidence and severity of PONV 48 hours after the surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Sun-Joon Bai, MD, Ph.D, Principal Investigator — Severance Hospital
Locations (1):
- Severance Hospital, Seoul, South Korea